CLINICAL TRIAL: NCT00431327
Title: Peer Coach Intervention to Improve Attendance to Scheduled Colonoscopy
Brief Title: Facilitators to Keeping Colonoscopy Appointments
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 705823
Record Dates: First submitted 2007-02-01; First posted 2007-02-05 (Estimated); Last update posted 2023-05-24 (Actual); Status verified 2023-05

CONDITIONS: Healthy
Keywords: patient navigator; peer support; colonoscopy; adherence; None: have to be scheduled for screening or diagnostic colonoscopy

INTERVENTIONS:
Behavioral: Peer coach phone call

SUMMARY:
To identify patients at risk for nonattendance to their first scheduled colonoscopy and to conduct a randomized trial of a theory-based, peer coach intervention on completing the scheduled colonoscopy.

DETAILED DESCRIPTION:
The potential to reduce the morbidity and mortality from colorectal cancer, the second most common cause of cancer death in the U.S. has been compromised because only about half of eligible patients have been appropriately screened. Patients contribute to inadequate colorectal cancer screening by failing to complete ordered tests. Several studies have reported low rates of attendance to scheduled sigmoidoscopy and colonoscopy studies. Because physicians offer limited counseling when ordering these tests, approaches are needed to address patient concerns and to promote adherence to scheduled colon studies. Therefore, we conducted a trial of a theory-based telephone intervention by patient 'peer coach' who was trained to address barriers to colonoscopy attendance versus a mailed professional brochure. The support was targeted to those at greatest risk of non-attendance.

ELIGIBILITY:
Inclusion Criteria:

* Age 50
* No prior colonoscopy in our health system records
* Patient in one of four primary care clinics within the University of Pennsylvania Health System
* Attended <75 of their primary care physicians visits within the past year

Exclusion Criteria:

* Colonoscopy not ordered by a primary care physician in a study clinic
* High readiness for the procedure
* A health care professional
* Had a prior colonoscopy outside of our health care system

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140
Dates: Start 2005-02; Study Completion 2006-10

PRIMARY OUTCOMES:
Attending the colonoscopy

CONTACTS AND LOCATIONS:
Overall Officials: Barbara J Turner, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States